CLINICAL TRIAL: NCT00622128
Title: Preventing Aggressive Behavior in Demented Patients
Acronym: PAVeD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Kunik, Mark - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MIRECC003
Record Dates: First submitted 2008-02-05; First posted 2008-02-22 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Dementia; Aggression
Keywords: Behavioral Research; Dementia; Aggression
MeSH Terms: conditions — Dementia; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Pilot study. Developing intervention
  Interventions: Behavioral: Preventing Aggressive Behavior in Demented Patients

INTERVENTIONS:
Behavioral: Preventing Aggressive Behavior in Demented Patients — Preventing Aggressive Behavior in Demented Patients

SUMMARY:
The purpose of this study is to develop and pilot test and non-pharmacological intervention designed to prevent the occurence of aggression in persons with dementia.

DETAILED DESCRIPTION:
An expert panel has met to review the investigators' prior work and literature to help create a non-pharmacological intervention designed to prevent the incidence of aggression. The investigators have created a manual based on prior work and expert input. Recruitment for pilot patients is now ready to begin. The purpose of the pilot will be to further adapt the intervention, assess feasibility, and examine recruitment options.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dementia,
* caregiver

Exclusion Criteria:

* history of aggression,
* residence of nursing homes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Aggression prevention | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Kunik, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States